CLINICAL TRIAL: NCT06386913
Title: Implementation and Evaluation of Measurement-Based Care Training
Brief Title: Implementation and Evaluation of Measurement-Based Care (MBC) Training
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Carilion Clinic (Other)
Collaborators: Virginia Polytechnic Institute and State University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: IRB-20-1065
Record Dates: First submitted 2024-04-15; First posted 2024-04-26 (Actual); Last update posted 2025-03-11 (Actual); Status verified 2025-03

CONDITIONS: Healthy
Keywords: Measurement-Based Care Training

STUDY DESIGN:
Intervention Model Description: Clinicians completed pre- and post-training surveys. Patient satisfaction was assessed prior to and after clinician training.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Clinician (Experimental): Mental health providers at Carilion Clinic completed Measurement-Base Care (MBC) training
  Interventions: Other: Training

INTERVENTIONS:
Other: Training — Measurement-Based Care Training

SUMMARY:
The purpose of this study is to get feedback on a new standardized Measurement-Based Care (MBC) provider training program.

DETAILED DESCRIPTION:
Measurement-Based Care (MBC) is the systematic ongoing collaborative evaluation of patient symptoms and well-being to inform clinical decision-making and behavioral health treatment. In this study, the goal is to receive feedback through surveys with experienced clinicians/practitioners to improve the training program design. Patient Satisfaction Surveys (PSS) were completed prior to and after clinician training. PSS assessed how Patient-Rated Outcome Measures (PROMs) are utilized by their clinicians, communicated during sessions and the ease to which completion is attainable as well as the patients' opinion regarding the use of such measures in treatment.

ELIGIBILITY:
Inclusion Criteria:

* Mental health providers in Carilion Clinic

Exclusion Criteria:

* None

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 56 (Actual)
Dates: Start 2021-02-09 (Actual); Primary Completion 2024-07-01 (Actual); Study Completion 2024-12-31 (Actual)

PRIMARY OUTCOMES:
Digital MBC training rate | 1 year
  Number of mental health providers who completed training out of the number providers invited
Assessing feasibility of a novel digital MBC training in mental health providers (FIM) | 1 year
  4-item questionnaire designed to assess implementation success by targeting an intervention feasibility
Assessing acceptability of a novel digital MBC training program in mental health providers (AIM) | 1 year
  4-item questionnaire designed to assess implementation success by targeting an intervention's acceptability
Assessing appropriateness of a novel digital MBC training program in mental health providers (IAM) | 1 year
  4-item questionnaire designed to assess implementation success by targeting an intervention's appropriateness

OTHER OUTCOMES:
Monitoring and Feedback Attitudes Scale (MFA) | 1 year
  14-item assessment of clinician belief regarding the potential benefits and risks of MBC
Attitudes Towards Standardized Assessment Scales: Monitoring and Feedback (ASA-MF) | 1 year
  18-item measurement of clinician attitudes toward using specific standardized measures and symptom monitoring to make clinical treatment decisions
Clinician Attitude and Satisfaction Survey (CASS) | 1 year
  7-item survey created to assess clinician attitudes of MBC

CONTACTS AND LOCATIONS:
Overall Officials: Robert L Trestman, PHD, MD, Study Director — Carilion Clinic
Locations (1):
- Carilion Clinic, Roanoke, Virginia, United States

IPD SHARING:
Plan to Share IPD: No